CLINICAL TRIAL: NCT05469776
Title: Retention of Both Cruciate Ligaments During Total Knee Arthroplasty: a Prospective Randomized Study
Brief Title: Bicruciate-retaining (2C) Total Knee Arthroplasty (TKA) Versus Posterior-stabilized (PS) Total Knee Arthroplasty (TKA)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Frédéric Lavoie, Orthopedic surgeon, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10.068
Record Dates: First submitted 2022-07-07; First posted 2022-07-22 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Total Knee Arthroplasty; Knee Osteoarthritis
Keywords: bicruciate-retaining; posterior-stabilized; Total Knee Arthroplasty; Knee Osteoarthritis; kinematic
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bicruciate-retaining total knee arthroplasty (Experimental): The prosthesis is minimally constrained and allows the preservation of both cruciate ligaments. All implants are cemented.
  Interventions: Procedure: bicruciate-retaining total knee arthroplasty
- posterior-stabilized total knee arthroplasty (Active Comparator): The prosthesis requires the excision of both cruciate ligaments
  Interventions: Procedure: posterior-stabilized total knee arthroplasty

INTERVENTIONS:
Procedure: bicruciate-retaining total knee arthroplasty
  Arms: bicruciate-retaining total knee arthroplasty
Procedure: posterior-stabilized total knee arthroplasty
  Arms: posterior-stabilized total knee arthroplasty

SUMMARY:
Total knee arthroplasty (TKA) with the sacrifice of the anterior cruciate ligament is the standard treatment for severe knee osteoarthritis. A number of studies on the kinematics of the prosthetic knee tend to show that implants that preserve the cruciate ligaments best reproduce the kinematics of the healthy knee. The goal is to compare the clinical and radiological results in patients undergoing total knee replacement surgery according to the type of prosthesis used. It is anticipated that the bicruciate-retaining prosthesis will result in better function of the operated knee than the posterior-stabilized prosthesis.

Method:

* Randomized controlled trial
* Monocentric
* Randomization will be done using sealed envelopes

DETAILED DESCRIPTION:
Posterior cruciate ligament replacement knee prostheses or posterior-stabilized (PS) are the most used type of prosthesis. Various studies of the kinematics of the prosthetic knee tend to show that implants that preserve both cruciate ligaments best reproduce the kinematics of the healthy knee. These implants are the unicondylar knee Arthroplasty - in which only one side of the femorotibial joint is replaced; most often the medial side - and the bicruciate-retaining total knee arthroplasty (BCR). The BCR prosthesis is perceived as technically difficult to install and has never been a great commercial success despite the scientific demonstration of its virtues for knee kinematics. Given the current trend among prosthetic implant manufacturers to optimize the performance of knee prostheses for younger, active patients, the retention of both cruciate ligaments appears to be an interesting alternative. Unfortunately, there are no good studies comparing the results of the BCR prosthesis to the PS prosthesis.

The goal is to compare the clinical and radiological results in patients undergoing total knee replacement surgery according to the type of prosthesis used (BCR vs PS).

The hypothesis is that the BCR prosthesis will result in better function of the operated knee than the PS prosthesis, resulting in joint kinematics closer to a healthy knee, better clinical scores and a higher activity level.

60 patients undergoing a total knee arthroplasty will be recruited. Randomization will be done intraoperatively using sealed envelopes once the indication for BCR TKA has been definitively established. Demographic data, medical history, clinical assessment and 4 questionnaires (IKS, KOOS, Marx and SF-12) will be completed prior to surgery. A standard x-ray, EOS imaging, TELOS radiological laximetry and a non-invasive evaluation of the 3D kinematics will be performed before the surgery.

Patients will complete the 4 questionnaires at 6 weeks, 6 months, 1 year, 2 years, 5 years and 10 years post-surgery. A standard radiological examination will be performed at the same follow-ups. TELOS radiological laximetry, EOS imaging and 3D kinematics assessment will be repeated at the 1-year follow-up post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients awaiting a total knee replacement who are candidates for a bi-cruciate retaining prosthesis
* Disabling bicompartmental gonarthrosis with failure of conservative treatment
* 70 years of age or younger at the time of the pre-operative consultation
* Intact and functional cruciate ligaments
* Coronal knee malalignment of 10 degrees or less
* Adequate preoperative range of motion, defined as maximum flexum (inability to fully extend the knee) of 10 degrees and flexion greater than 90 degrees
* Adequate intraoperative knee exposure to allow preservation of both cruciate ligaments

Exclusion Criteria:

* Inability to undergo an EOS examination, defined as the inability to stand or morbid obesity (inability of the patient to enter the EOS machine, which is relatively cramped)
* Inability to walk on a treadmill and squat
* Pregnant women to avoid unnecessary fetal radiation
* Illiteracy, language barrier and any other reason that prevents patients from answering the questionnaires

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in KOOS pain score | Change from baseline (pre surgery) KOOS pain score at 10 years after the surgery
  KOOS pain score; 0-100 scale, 0: extreme problems 100: no problems

SECONDARY OUTCOMES:
Change in KOOS pain score | Change from baseline (pre surgery) KOOS pain score at 6 weeks after the surgery
  KOOS pain score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS pain score | Change from baseline (pre surgery) KOOS pain score at 6 months after the surgery
  KOOS pain score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS pain score | Change from baseline (pre surgery) KOOS pain score at 1 year after the surgery
  KOOS pain score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS pain score | Change from baseline (pre surgery) KOOS pain score at 2 years after the surgery
  KOOS pain score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS pain score | Change from baseline (pre surgery) KOOS pain score at 5 years after the surgery
  KOOS pain score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS symptoms score | Change from baseline (pre surgery) KOOS pain symptoms at 6 weeks after the surgery
  KOOS symptoms score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS symptoms score | Change from baseline (pre surgery) KOOS symptoms score at 6 months after the surgery
  KOOS symptoms score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS symptoms score | Change from baseline (pre surgery) KOOS symptoms score at 1 year after the surgery
  KOOS symptoms score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS symptoms score | Change from baseline (pre surgery) KOOS symptoms score at 2 years after the surgery
  KOOS symptoms score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS symptoms score | Change from baseline (pre surgery) KOOS pain symptoms at 5 years after the surgery
  KOOS symptoms score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS symptoms score | Change from baseline (pre surgery) KOOS pain symptoms at 10 years after the surgery
  KOOS symptoms score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS activity of daily living score | Change from baseline (pre surgery) KOOS activity of daily living at 6 weeks after the surgery
  KOOS symptoms score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS activity of daily living score | Change from baseline (pre surgery) KOOS activity of daily living score at 6 months after the surgery
  KOOS activity of daily living score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS activity of daily living score | Change from baseline (pre surgery) KOOS activity of daily living score at 1 year after the surgery
  KOOS activity of daily living score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS activity of daily living score | Change from baseline (pre surgery) KOOS activity of daily living score at 2 years after the surgery
  KOOS activity of daily living score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS activity of daily living score | Change from baseline (pre surgery) KOOS activity of daily living at 5 years after the surgery
  KOOS symptoms score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS activity of daily living score | Change from baseline (pre surgery) KOOS activity of daily living at 10 years after the surgery
  KOOS symptoms score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS sport and recreation score | Change from baseline (pre surgery) KOOS sport and recreation at 6 weeks after the surgery
  KOOS sport and recreation score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS sport and recreation score | Change from baseline (pre surgery) KOOS sport and recreation score at 6 months after the surgery
  KOOS sport and recreation score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS sport and recreation score | Change from baseline (pre surgery) KOOS sport and recreation score at 1 year after the surgery
  KOOS sport and recreation score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS sport and recreation score | Change from baseline (pre surgery) KOOS sport and recreation score at 2 years after the surgery
  KOOS sport and recreation score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS sport and recreation score | Change from baseline (pre surgery) KOOS sport and recreation at 5 years after the surgery
  KOOS sport and recreation score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS sport and recreation score | Change from baseline (pre surgery) KOOS sport and recreation at 10 years after the surgery
  KOOS sport and recreation score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS quality of life score | Change from baseline (pre surgery) KOOS quality of life at 6 weeks after the surgery
  KOOS quality of life score score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS quality of life score | Change from baseline (pre surgery) KOOS quality of life score at 6 months after the surgery
  KOOS quality of life score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS quality of life score | Change from baseline (pre surgery) KOOS quality of life score at 1 year after the surgery
  KOOS quality of life score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS quality of life score | Change from baseline (pre surgery) KOOS quality of life score at 2 years after the surgery
  KOOS quality of life score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS quality of life score | Change from baseline (pre surgery) KOOS quality of life at 5 years after the surgery
  KOOS quality of life score; 0-100 scale, 0: extreme problems 100: no problems
Change in KOOS quality of life score | Change from baseline (pre surgery) KOOS quality of life at 10 years after the surgery
  KOOS quality of life score; 0-100 scale, 0: extreme problems 100: no problems
Change in MARX score | Change from baseline (pre surgery) MARX score at 6 weeks after the surgery
  MARX activity rating scale; 0-16, 0: less frequent sport participation 16: more frequent sport participation
Change in MARX score | Change from baseline (pre surgery) MARX score at 6 months after the surgery
  MARX activity rating scale; 0-16, 0: less frequent sport participation 16: more frequent sport participation
Change in MARX score | Change from baseline (pre surgery) MARX score at 1 year after the surgery
  MARX activity rating scale; 0-16, 0: less frequent sport participation 16: more frequent sport participation
Change in MARX score | Change from baseline (pre surgery) MARX score at 2 years after the surgery
  MARX activity rating scale; 0-16, 0: less frequent sport participation 16: more frequent sport participation
Change in MARX score | Change from baseline (pre surgery) MARX score at 5 yearss after the surgery
  MARX activity rating scale; 0-16, 0: less frequent sport participation 16: more frequent sport participation
Change in MARX score | Change from baseline (pre surgery) MARX score at 10 yearss after the surgery
  MARX activity rating scale; 0-16, 0: less frequent sport participation 16: more frequent sport participation
Change in International Knee Society scoring system (IKS) : knee score | Change from baseline (pre surgery) IKS Knee score at 6 weeks after the surgery
  IKS Knee score; 0-100, 0: poor condition of the knee 100: better condition of the knee
Change in International Knee Society scoring system (IKS) : knee score | Change from baseline (pre surgery) IKS Knee score at 6 months after the surgery
  IKS Knee score; 0-100, 0: poor condition of the knee 100: better condition of the knee
Change in International Knee Society scoring system (IKS) : knee score | Change from baseline (pre surgery) IKS Knee score at 1 year after the surgery
  IKS Knee score; 0-100, 0: poor condition of the knee 100: better condition of the knee
Change in International Knee Society scoring system (IKS) : knee score | Change from baseline (pre surgery) IKS Knee score at 2 years after the surgery
  IKS Knee score; 0-100, 0: poor condition of the knee 100: better condition of the knee
Change in International Knee Society scoring system (IKS) : knee score | Change from baseline (pre surgery) IKS Knee score at 5 years after the surgery
  IKS Knee score; 0-100, 0: poor condition of the knee 100: better condition of the knee
Change in International Knee Society scoring system (IKS) : knee score | Change from baseline (pre surgery) IKS Knee score at 10 years after the surgery
  IKS Knee score; 0-100, 0: poor condition of the knee 100: better condition of the knee
Change in International Knee Society scoring system (IKS) : function score | Change from baseline (pre surgery) IKS function score at 6 weeks after the surgery
  IKS Knee score; 0-100, 0: severe functional disability 100: no disability
Change in International Knee Society scoring system (IKS) : function score | Change from baseline (pre surgery) IKS function score at 6 months after the surgery
  IKS Knee score; 0-100, 0: severe functional disability 100: no disability
Change in International Knee Society scoring system (IKS) : function score | Change from baseline (pre surgery) IKS function score at 1 year after the surgery
  IKS Knee score; 0-100, 0: severe functional disability 100: no disability
Change in International Knee Society scoring system (IKS) : function score | Change from baseline (pre surgery) IKS function score at 2 years after the surgery
  IKS Knee score; 0-100, 0: severe functional disability 100: no disability
Change in International Knee Society scoring system (IKS) : function score | Change from baseline (pre surgery) IKS function score at 5 years after the surgery
  IKS Knee score; 0-100, 0: severe functional disability 100: no disability
Change in International Knee Society scoring system (IKS) : function score | Change from baseline (pre surgery) IKS function score at 10 years after the surgery
  IKS Knee score; 0-100, 0: severe functional disability 100: no disability
Change in Knee Range of Motion (ROM) | Change from baseline (pre surgery) ROM at 6 weeks after the surgery
  Genu Recurvatum, Genu Flexum and Knee maximal flexion, angle in degrees ranging from 0 to 160
Change in Knee Range of Motion (ROM) | Change from baseline (pre surgery) ROM at 6 months after the surgery
  Genu Recurvatum, Genu Flexum and Knee maximal flexion, angle in degrees ranging from 0 to 160
Change in Knee Range of Motion (ROM) | Change from baseline (pre surgery) ROM at 1 year after the surgery
  Genu Recurvatum, Genu Flexum and Knee maximal flexion, angle in degrees ranging from 0 to 160
Change in Knee Range of Motion (ROM) | Change from baseline (pre surgery) ROM at 2 years after the surgery
  Genu Recurvatum, Genu Flexum and Knee maximal flexion, angle in degrees ranging from 0 to 160
Change in Knee Range of Motion (ROM) | Change from baseline (pre surgery) ROM at 5 years after the surgery
  Genu Recurvatum, Genu Flexum and Knee maximal flexion, angle in degrees ranging from 0 to 160
Change in Knee Range of Motion (ROM) | Change from baseline (pre surgery) ROM at 10 years after the surgery
  Genu Recurvatum, Genu Flexum and Knee maximal flexion, angle in degrees ranging from 0 to 160
Change in Lower limb morphology in the coronal plane | Change from baseline (pre surgery) Lower limb morphology in the coronal plane at 6 weeks after the surgery
  Lower limb morphology in the coronal plane; neutral: 176-184 degrees varus: <176 degrees valgus: > 184 degrees
Change in Lower limb morphology in the coronal plane | Change from baseline (pre surgery) Lower limb morphology in the coronal plane at 6 months after the surgery
  Lower limb morphology in the coronal plane; neutral: 176-184 degrees varus: <176 degrees valgus: > 184 degrees
Change in Lower limb morphology in the coronal plane | Change from baseline (pre surgery) Lower limb morphology in the coronal plane at 1 year after the surgery
  Lower limb morphology in the coronal plane; neutral: 176-184 degrees varus: <176 degrees valgus: > 184 degrees
Change in Lower limb morphology in the coronal plane | Change from baseline (pre surgery) Lower limb morphology in the coronal plane at 2 years after the surgery
  Lower limb morphology in the coronal plane; neutral: 176-184 degrees varus: <176 degrees valgus: > 184 degrees
Change in Lower limb morphology in the coronal plane | Change from baseline (pre surgery) Lower limb morphology in the coronal plane at 5 years after the surgery
  Lower limb morphology in the coronal plane; neutral: 176-184 degrees varus: <176 degrees valgus: > 184 degrees
Change in Lower limb morphology in the coronal plane | Change from baseline (pre surgery) Lower limb morphology in the coronal plane at 10 years after the surgery
  Lower limb morphology in the coronal plane; neutral: 176-184 degrees varus: <176 degrees valgus: > 184 degrees
Change in Knee alignment : Hip-knee-ankle (HKA) | Change from baseline (pre surgery) HKA at 6 weeks after the surgery
  Hip-knee-ankle (HKA); 150-210 degrees
Change in Knee alignment : Hip-knee-ankle (HKA) | Change from baseline (pre surgery) HKA at 6 months after the surgery
  Hip-knee-ankle (HKA); 150-210 degrees
Change in Knee alignment : Hip-knee-ankle (HKA) | Change from baseline (pre surgery) HKA at 1 year after the surgery
  Hip-knee-ankle (HKA); 150-210 degrees
Change in Knee alignment : Hip-knee-ankle (HKA) | Change from baseline (pre surgery) HKA at 2 years after the surgery
  Hip-knee-ankle (HKA); 150-210 degrees
Change in Knee alignment : Hip-knee-ankle (HKA) | Change from baseline (pre surgery) HKA at 5 years after the surgery
  Hip-knee-ankle (HKA); 150-210 degrees
Change in Knee alignment : Hip-knee-ankle (HKA) | Change from baseline (pre surgery) HKA at 10 years after the surgery
  Hip-knee-ankle (HKA); 150-210 degrees
Change in Knee alignment : Hip-knee-shaft (HKS) | Change from baseline (pre surgery) HKS at 6 weeks after the surgery
  Hip-knee-shaft (HKS); 2-15 degrees
Change in Knee alignment : Hip-knee-shaft (HKS) | Change from baseline (pre surgery) HKS at 6 months after the surgery
  Hip-knee-shaft (HKS); 2-15 degrees
Change in Knee alignment : Hip-knee-shaft (HKS) | Change from baseline (pre surgery) HKS at 1 year after the surgery
  Hip-knee-shaft (HKS); 2-15 degrees
Change in Knee alignment : Hip-knee-shaft (HKS) | Change from baseline (pre surgery) HKS at 2 years after the surgery
  Hip-knee-shaft (HKS); 2-15 degrees
Change in Knee alignment : Hip-knee-shaft (HKS) | Change from baseline (pre surgery) HKS at 5 years after the surgery
  Hip-knee-shaft (HKS); 2-15 degrees
Change in Knee alignment : Hip-knee-shaft (HKS) | Change from baseline (pre surgery) HKS at 10 years after the surgery
  Hip-knee-shaft (HKS); 2-15 degrees
Change in Knee alignment : Medial distal femoral angle (MDFA) | Change from baseline (pre surgery) MDFA at 6 weeks after the surgery
  Medial distal femoral angle (MDFA); 75-100 degrees
Change in Knee alignment : Medial distal femoral angle (MDFA) | Change from baseline (pre surgery) MDFA at 6 months after the surgery
  Medial distal femoral angle (MDFA); 75-100 degrees
Change in Knee alignment : Medial distal femoral angle (MDFA) | Change from baseline (pre surgery) MDFA at 1 year after the surgery
  Medial distal femoral angle (MDFA); 75-100 degrees
Change in Knee alignment : Medial distal femoral angle (MDFA) | Change from baseline (pre surgery) MDFA at 2 years after the surgery
  Medial distal femoral angle (MDFA); 75-100 degrees
Change in Knee alignment : Medial distal femoral angle (MDFA) | Change from baseline (pre surgery) MDFA at 5 years after the surgery
  Medial distal femoral angle (MDFA); 75-100 degrees
Change in Knee alignment : Medial distal femoral angle (MDFA) | Change from baseline (pre surgery) MDFA at 10 years after the surgery
  Medial distal femoral angle (MDFA); 75-100 degrees
Change in Knee alignment : Medial proximal tibial angle (MPTA) | Change from baseline (pre surgery) MPTA at 6 weeks after the surgery
  Medial proximal tibial angle (MPTA); 70-110 degrees
Change in Knee alignment : Medial proximal tibial angle (MPTA) | Change from baseline (pre surgery) MPTA at 6 months after the surgery
  Medial proximal tibial angle (MPTA); 70-110 degrees
Change in Knee alignment : Medial proximal tibial angle (MPTA) | Change from baseline (pre surgery) MPTA at 1 year after the surgery
  Medial proximal tibial angle (MPTA); 70-110 degrees
Change in Knee alignment : Medial proximal tibial angle (MPTA) | Change from baseline (pre surgery) MPTA at 2 years after the surgery
  Medial proximal tibial angle (MPTA); 70-110 degrees
Change in Knee alignment : Medial proximal tibial angle (MPTA) | Change from baseline (pre surgery) MPTA at 5 years after the surgery
  Medial proximal tibial angle (MPTA); 70-110 degrees
Change in Knee alignment : Medial proximal tibial angle (MPTA) | Change from baseline (pre surgery) MPTA at 10 years after the surgery
  Medial proximal tibial angle (MPTA); 70-110 degrees
Change in Knee ligament laxity : Anterior/Posterior Instability | Change from baseline (pre surgery) Anterior/Posterior Instability at 6 weeks after the surgery
  Anterior/Posterior Instability; measured at 90 degrees; none, moderate < 5mm, severe >5 mm
Change in Knee ligament laxity : Anterior/Posterior Instability | Change from baseline (pre surgery) Anterior/Posterior Instability at 6 months after the surgery
  Anterior/Posterior Instability; measured at 90 degrees; none, moderate < 5mm, severe >5 mm
Change in Knee ligament laxity : Anterior/Posterior Instability | Change from baseline (pre surgery) Anterior/Posterior Instability at 1 year after the surgery
  Anterior/Posterior Instability; measured at 90 degrees; none, moderate < 5mm, severe >5 mm
Change in Knee ligament laxity : Anterior/Posterior Instability | Change from baseline (pre surgery) Anterior/Posterior Instability at 2 years after the surgery
  Anterior/Posterior Instability; measured at 90 degrees; none, moderate < 5mm, severe >5 mm
Change in Knee ligament laxity : Anterior/Posterior Instability | Change from baseline (pre surgery) Anterior/Posterior Instability at 5 years after the surgery
  Anterior/Posterior Instability; measured at 90 degrees; none, moderate < 5mm, severe >5 mm
Change in Knee ligament laxity : Anterior/Posterior Instability | Change from baseline (pre surgery) Anterior/Posterior Instability at 10 years after the surgery
  Anterior/Posterior Instability; measured at 90 degrees; none, moderate < 5mm, severe >5 mm
Change in Knee ligament laxity : Medial/Lateral Instability | Change from baseline (pre surgery) Medial/Lateral Instability at 6 weeks after the surgery
  Medial/Lateral Instability; measured in full extension; none, little < 5 mm, moderate = 5mm, severe > 5 mm
Change in Knee ligament laxity : Medial/Lateral Instability | Change from baseline (pre surgery) Medial/Lateral Instability at 6 months after the surgery
  Medial/Lateral Instability; measured in full extension; none, little < 5 mm, moderate = 5mm, severe > 5 mm
Change in Knee ligament laxity : Medial/Lateral Instability | Change from baseline (pre surgery) Medial/Lateral Instability at 1 year after the surgery
  Medial/Lateral Instability; measured in full extension; none, little < 5 mm, moderate = 5mm, severe > 5 mm
Change in Knee ligament laxity : Medial/Lateral Instability | Change from baseline (pre surgery) Medial/Lateral Instability at 2 years after the surgery
  Medial/Lateral Instability; measured in full extension; none, little < 5 mm, moderate = 5mm, severe > 5 mm
Change in Knee ligament laxity : Medial/Lateral Instability | Change from baseline (pre surgery) Medial/Lateral Instability at 5 years after the surgery
  Medial/Lateral Instability; measured in full extension; none, little < 5 mm, moderate = 5mm, severe > 5 mm
Change in Knee ligament laxity : Medial/Lateral Instability | Change from baseline (pre surgery) Medial/Lateral Instability at 10 years after the surgery
  Medial/Lateral Instability; measured in full extension; none, little < 5 mm, moderate = 5mm, severe > 5 mm
Change in Patellar apprehension test | Change from baseline (pre surgery) Patellofemoral Instability at 6 weeks after the surgery
  Clinical physical examination for patellofemoral instability; Patellar apprehension test; normal, apprehension, apprehension and dislocation
Change in Patellar apprehension test | Change from baseline (pre surgery) Patellofemoral Instability at 6 months after the surgery
  Clinical physical examination for patellofemoral instability; Patellar apprehension test; normal, apprehension, apprehension and dislocation
Change in Patellar apprehension test | Change from baseline (pre surgery) Patellofemoral Instability at 1 year after the surgery
  Clinical physical examination for patellofemoral instability; Patellar apprehension test; normal, apprehension, apprehension and dislocation
Change in Patellar apprehension test | Change from baseline (pre surgery) Patellofemoral Instability at 2 years after the surgery
  Clinical physical examination for patellofemoral instability; Patellar apprehension test; normal, apprehension, apprehension and dislocation
Change in Patellar apprehension test | Change from baseline (pre surgery) Patellofemoral Instability at 5 years after the surgery
  Clinical physical examination for patellofemoral instability; Patellar apprehension test; normal, apprehension, apprehension and dislocation
Change in Patellar apprehension test | Change from baseline (pre surgery) Patellofemoral Instability at 10 years after the surgery
  Clinical physical examination for patellofemoral instability; Patellar apprehension test; normal, apprehension, apprehension and dislocation
Change in Physical Activity Level Scale | Change from baseline (pre surgery) Physical Activity Level at 6 weeks after the surgery
  Physical Activity Level Scale; None, Mild, Moderate, Strenuous, Competitive
Change in Physical Activity Level Scale | Change from baseline (pre surgery) Physical Activity Level at 6 months after the surgery
  Physical Activity Level Scale; None, Mild, Moderate, Strenuous, Competitive
Change in Physical Activity Level Scale | Change from baseline (pre surgery) Physical Activity Level at 1 year after the surgery
  Physical Activity Level Scale; None, Mild, Moderate, Strenuous, Competitive
Change in Physical Activity Level Scale | Change from baseline (pre surgery) Physical Activity Level at 2 years after the surgery
  Physical Activity Level Scale; None, Mild, Moderate, Strenuous, Competitive
Change in Physical Activity Level Scale | Change from baseline (pre surgery) Physical Activity Level at 5 years after the surgery
  Physical Activity Level Scale; None, Mild, Moderate, Strenuous, Competitive
Change in Physical Activity Level Scale | Change from baseline (pre surgery) Physical Activity Level at 10 years after the surgery
  Physical Activity Level Scale; None, Mild, Moderate, Strenuous, Competitive
Change in Physical Activities Scale | Change from baseline (pre surgery) Physical Activities at 6 weeks after the surgery
  Physical Activities Scale; Sedentary / very little, Physical work, Aerobic, Sport(s) without pivot, Sport(s) with pivot
Change in Physical Activities Scale | Change from baseline (pre surgery) Physical Activities at 6 months after the surgery
  Physical Activities Scale; Sedentary / very little, Physical work, Aerobic, Sport(s) without pivot, Sport(s) with pivot
Change in Physical Activities Scale | Change from baseline (pre surgery) Physical Activities at 1 year after the surgery
  Physical Activities Scale; Sedentary / very little, Physical work, Aerobic, Sport(s) without pivot, Sport(s) with pivot
Change in Physical Activities Scale | Change from baseline (pre surgery) Physical Activities at 2 years after the surgery
  Physical Activities Scale; Sedentary / very little, Physical work, Aerobic, Sport(s) without pivot, Sport(s) with pivot
Change in Physical Activities Scale | Change from baseline (pre surgery) Physical Activities at 5 years after the surgery
  Physical Activities Scale; Sedentary / very little, Physical work, Aerobic, Sport(s) without pivot, Sport(s) with pivot
Change in Physical Activities Scale | Change from baseline (pre surgery) Physical Activities at 10 years after the surgery
  Physical Activities Scale; Sedentary / very little, Physical work, Aerobic, Sport(s) without pivot, Sport(s) with pivot
Change in 12-Item Short Form Survey (SF-12) score | Change from baseline (pre surgery) SF-12 Questionnaire at 6 weeks after the surgery
  SF-12; Physical component summary (PCS-12), Mental component summary (MCS-12), the scores are reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average.
Change in 12-Item Short Form Survey (SF-12) score | Change from baseline (pre surgery) SF-12 Questionnaire at 6 months after the surgery
  SF-12; Physical component summary (PCS-12), Mental component summary (MCS-12), the scores are reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average.
Change in 12-Item Short Form Survey (SF-12) score | Change from baseline (pre surgery) SF-12 Questionnaire at 1 year after the surgery
  SF-12; Physical component summary (PCS-12), Mental component summary (MCS-12), the scores are reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average.
Change in 12-Item Short Form Survey (SF-12) score | Change from baseline (pre surgery) SF-12 Questionnaire at 2 years after the surgery
  SF-12; Physical component summary (PCS-12), Mental component summary (MCS-12), the scores are reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average.
Change in 12-Item Short Form Survey (SF-12) score | Change from baseline (pre surgery) SF-12 Questionnaire at 5 years after the surgery
  SF-12; Physical component summary (PCS-12), Mental component summary (MCS-12), the scores are reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average.
Change in 12-Item Short Form Survey (SF-12) score | Change from baseline (pre surgery) SF-12 Questionnaire at 10 years after the surgery
  SF-12; Physical component summary (PCS-12), Mental component summary (MCS-12), the scores are reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS-12 and MCS-12 are both 50 points. The United States population standard deviation is 10 points. So each 10 increment of 10 points above or below 50, corresponds to one standard deviation away from the average.
Change in TELOS radiological laximetry | Change from baseline (pre surgery) TELOS radiological laximetry at 1 year after the surgery
  TELOS radiological laximetry of both knees; varus and valgus laxity with knees in extension, anterior-posterior laxity of the knees at 20 and 90 degrees of flexion
Change in EOS imaging pseudo-kinematic - standardized squatting task - knee flexion and extension | Change from baseline (pre surgery) EOS imaging pseudo-kinematic at 1 year after the surgery
  EOS imaging of both knees during a standardized squatting task; knee rotation around the media-lateral axis (knee flexion and extension), degrees
Change in EOS imaging pseudo-kinematic - standardized squatting task - knee abduction and adduction | Change from baseline (pre surgery) EOS imaging pseudo-kinematic at 1 year after the surgery
  EOS imaging of both knees during a standardized squatting task; knee rotation around the anteroposterior axis (knee abduction and adduction), degrees
Change in EOS imaging pseudo-kinematic - standardized squatting task - knee internal and external rotation | Change from baseline (pre surgery) EOS imaging pseudo-kinematic at 1 year after the surgery
  EOS imaging of both knees during a standardized squatting task; knee rotation around the longitudinal axis (knee internal and external rotation), degrees
Change in EOS imaging pseudo-kinematic - free squatting task - knee flexion and extension | Change from baseline (pre surgery) EOS imaging pseudo-kinematic at 1 year after the surgery
  EOS imaging of both knees during a free squatting task; knee rotation around the media-lateral axis (knee flexion and extension), degrees
Change in EOS imaging pseudo-kinematic - free squatting task - knee abduction and adduction | Change from baseline (pre surgery) EOS imaging pseudo-kinematic at 1 year after the surgery
  EOS imaging of both knees during a free squatting task; knee rotation around the anteroposterior axis (knee abduction and adduction), degrees
Change in EOS imaging pseudo-kinematic - free squatting task - knee internal and external rotation | Change from baseline (pre surgery) EOS imaging pseudo-kinematic at 1 year after the surgery
  EOS imaging of both knees during a free squatting task; knee rotation around the longitudinal axis (knee internal and external rotation), degrees
Changes in 3D knee kinematics assessment during walking - knee flexion and extension | Change from baseline (pre surgery) 3D kinematics assessment at 1 year after the surgery
  3D kinematics assessment during walking, the knee kinematics will be assessed using the kneeKG system, knee rotation around the media-lateral axis (knee flexion and extension), degrees
Changes in 3D knee kinematics assessment during walking measured with the KneeKG system - knee abduction and adduction | Change from baseline (pre surgery) 3D kinematics assessment at 1 year after the surgery
  3D kinematics assessment during walking, the knee kinematics will be assessed using the kneeKG system, knee rotation around the anteroposterior axis (knee abduction and adduction), degrees
Changes in 3D knee kinematics assessment during walking measured with the KneeKG system - knee internal and external rotation | Change from baseline (pre surgery) 3D kinematics assessment at 1 year after the surgery
  3D kinematics assessment during walking, the knee kinematics will be assessed using the kneeKG system, knee rotation around the longitudinal axis (knee internal and external rotation), degrees

OTHER OUTCOMES:
Change in Body Mass Index (BMI) | Change from baseline (pre surgery) BMI at 6 weeks after the surgery
  BMI; <18.5->30, <18.5: underweight 18.5-24.9: normal weight 25.0-29.9: overweight >30.0: obesity
Change in Body Mass Index (BMI) | Change from baseline (pre surgery) BMI at 6 months after the surgery
  BMI; <18.5->30, <18.5: underweight 18.5-24.9: normal weight 25.0-29.9: overweight >30.0: obesity
Change in Body Mass Index (BMI) | Change from baseline (pre surgery) BMI at 1 year after the surgery
  BMI; <18.5->30, <18.5: underweight 18.5-24.9: normal weight 25.0-29.9: overweight >30.0: obesity
Change in Body Mass Index (BMI) | Change from baseline (pre surgery) BMI at 2 years after the surgery
  BMI; <18.5->30, <18.5: underweight 18.5-24.9: normal weight 25.0-29.9: overweight >30.0: obesity

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Lavoie, MD, M.Sc, Principal Investigator — CHUM
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cloutier JM. Long-term results after nonconstrained total knee arthroplasty. Clin Orthop Relat Res. 1991 Dec;(273):63-5. PMID 1959288
- [Background] Goutallier D, Manicom O, Van Driessche S. [Total knee arthroplasty with bicruciate preservation: Comparison versus the same posterostabilized design at eight years follow-up]. Rev Chir Orthop Reparatrice Appar Mot. 2008 Oct;94(6):585-95. doi: 10.1016/j.rco.2008.04.012. Epub 2008 Jul 11. French. PMID 18929754
- [Background] Goutallier D, Glorion C. [Critical assessment of the functional advantage of preserving the 2 cruciate ligaments in total knee prosthesis. Experience with the Hermes' prosthesis]. Acta Orthop Belg. 1991;57 Suppl 2:128-9. No abstract available. French. PMID 1792876
- [Background] Henckel J, Richards R, Lozhkin K, Harris S, Rodriguez y Baena FM, Barrett AR, Cobb JP. Very low-dose computed tomography for planning and outcome measurement in knee replacement. The imperial knee protocol. J Bone Joint Surg Br. 2006 Nov;88(11):1513-8. doi: 10.1302/0301-620X.88B11.17986. PMID 17075100
- [Background] Insall JN, Binazzi R, Soudry M, Mestriner LA. Total knee arthroplasty. Clin Orthop Relat Res. 1985 Jan-Feb;(192):13-22. PMID 3967412
- [Background] Insall JN, Dorr LD, Scott RD, Scott WN. Rationale of the Knee Society clinical rating system. Clin Orthop Relat Res. 1989 Nov;(248):13-4. PMID 2805470
- [Background] Komistek RD, Allain J, Anderson DT, Dennis DA, Goutallier D. In vivo kinematics for subjects with and without an anterior cruciate ligament. Clin Orthop Relat Res. 2002 Nov;(404):315-25. doi: 10.1097/00003086-200211000-00047. PMID 12439275
- [Background] Komistek RD, Scott RD, Dennis DA, Yasgur D, Anderson DT, Hajner ME. In vivo comparison of femorotibial contact positions for press-fit posterior stabilized and posterior cruciate-retaining total knee arthroplasties. J Arthroplasty. 2002 Feb;17(2):209-16. doi: 10.1054/arth.2002.29329. PMID 11847622
- [Background] Laskin RS. Choosing your implant: cemented, tricompartmental, and posterior stabilized. J Arthroplasty. 2005 Jun;20(4 Suppl 2):7-9. doi: 10.1016/j.arth.2005.03.012. PMID 15991119
- [Background] Lee SY, Matsui N, Kurosaka M, Komistek RD, Mahfouz M, Dennis DA, Yoshiya S. A posterior-stabilized total knee arthroplasty shows condylar lift-off during deep knee bends. Clin Orthop Relat Res. 2005 Jun;(435):181-4. doi: 10.1097/01.blo.0000155013.31327.dc. PMID 15930936
- [Background] van den Bekerom MP, Patt TW, Kleinhout MY, van der Vis HM, Albers GH. Early complications after high tibial osteotomy: a comparison of two techniques. J Knee Surg. 2008 Jan;21(1):68-74. doi: 10.1055/s-0030-1247797. PMID 18300676